CLINICAL TRIAL: NCT05486442
Title: Acceptance and Commitment Training for Weight-related Experiential Avoidance
Brief Title: ACT for Weight-related Experiential Avoidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahcesehir Cyprus University (Other)
Responsible Party: Principal Investigator, Buse Keskindag, Principal Investigator, Bahcesehir Cyprus University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NEU/SS/2022/1208
Record Dates: First submitted 2022-07-30; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group received ACT training in the group setting aiming to reduce weight-related experiential avoidance. This included 6 sessions in total. Each session was completed approximately in 80 mins.
  Interventions: Behavioral: ACT for weight-related experiential avoidance
- Control group (No Intervention): Participants in the control group did not receive any manipulation

INTERVENTIONS:
Behavioral: ACT for weight-related experiential avoidance — Participants in the experimental group received weight concern-related ACT training in a group setting. Each session focused on different dimensions of ACT and included relevant exercises and homeworks. Dimensions studied included creative hopelessness, control strategies, mindfulness exercises, values and barries to values and commitment to action.
  Arms: Experimental group

SUMMARY:
This study aimed to investigate whether Acceptance and Commitment Therapy/Training would be helpful to reduce weight-related experiential avoidance among individuals who reported weight concern

DETAILED DESCRIPTION:
This quasi-experimental study aimed to examine the efficacy of Acceptance and Commitment Therapy/Training (ACT) in reducing weight-related experiential avoidance. Data were collected with a convenience sampling technique. After obtaining ethical approval, participants were invited to participate in the study via advertisements, and online posts. Due to the small sample size, participants who were willing to attend group discussions were included in the experimental group. Participants in the control group did not receive manipulation. All participants were provided with an informed consent form. All participants completed a questionnaire measuring outcomes (weight-related experiential avoidance, general experiential avoidance, eating attitudes, and social physique anxiety) at pre-test, post-test, and follow-up. Participants in the experimental group received ACT training including 6 sessions. The protocol was adapted from Pearson et al. (2012) with their permission. Each session took approximately 80 mins. Several aspects of ACT approach were discussed in the sessions. In session one, ACT approach was introduced. In session two, creative hopelessness was discussed. In session three, control strategies related to weight concern were identified. In session four, mindfulness exercises were completed. In the fifth session, values for meaningful life experience were discussed. In the last, sixth session, the ways to commit to action were discussed. Each session included exercises and homework. At the end of the study, the participants were provided with debrief form.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were 18 years and older
* Ability to read and understand Turkish

Exclusion Criteria:

* Individuals who have received mental health intervention over the last one year
* and those who were diagnosed with an eating disorder were excluded from the analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Change in weight-related experiential avoidance | At three time points (pre-intervention [baseline], immediately after the intervention, and at three weeks after the intervention)
  It was measured by Acceptance and Action Questionnaire for Weight-Related Difficulties-Revised. The scale includes 10 items that are rated on 7 points scale (1 = not true at all - 7 = completely true). Higher scores indicate greater weight related experiential avoidance.

SECONDARY OUTCOMES:
Change in eating attitudes | At three time points (pre-intervention [baseline], immediately after the intervention, and at three weeks after the intervention)
  Eating attitudes were measured by The Eating Attitudes Test-26. It includes 26 items that are rated on 4 point scale ('3 = Always, 2 = Usually, 1 = Often, 0 = Sometimes, Rarely, and Never'). The last item (26) requires reverse coding. Scores 20 and above indicate dysfunctional eating attitudes.
Change in general experiential avoidance | At three time points (pre-intervention [baseline], immediately after the intervention, and at three weeks after the intervention)
  It was measured by Acceptance and Action Questionnaire-II. It includes 7 items that are rated on 7 point scale (1 = never true - 7 = always true). Minimum and maximum scores range between 7 and 49 points. Higher scores indicate greater general experiential avoidance (psychological inflexibility).
Change in social physique anxiety | At three time points (pre-intervention [baseline], immediately after the intervention, and at three weeks after the intervention)
  It was measured by The Social Physique Anxiety Scale. The scale includes 12 items are rated on a 5-point scale (1=not at all true to 5=extremely true). Higher scores indicate a higher level of anxiety related to the social physique. Only item 1, 2, 5, 8 and 11 requires reverse coding.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Karaaziz, PhD, Study Director — Near East University
Locations (1):
- Near East University, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearson, Adria N., Victoria M. Follette, and Steven C. Hayes.
- See also: Protocol of this study was adapted with permission of corresponding author — https://doi.org/10.1016/j.cbpra.2011.03.001